CLINICAL TRIAL: NCT06210763
Title: Inspiratory Muscle Training Outcomes in Sufferers of Severe Walking Disabilities and Intensive Care Unit Acquired Weakness
Brief Title: IMT Outcomes in Sufferers of Severe Walking Disabilities and Intensive Care Unit Acquired Weakness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Cardiovascular, Respiratory disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004624
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Intensive Care Unit Acquired Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): twenty ICU-acquired weakness elderly patients will receive chest physiotherapy (cough training, vibration, percussion, rib springing, and postural drainage), 30 minutes of resisted training on upper- and lower-limb muscles (15 min on upper limb and 15 min on lower limb), and 30 minutes of neuromuscular electrical stimulation of lower- and upper-limb muscles (triceps and wrist extensors, dorsiflexors, and quadriceps). sessions will be executed 5 times weekly). this Group will receive 3-set IMT (two sessions daily via threshold IMT, the set contain 10 repetitions) 5 times weekly. The study duration will be 1 month.
  Interventions: Behavioral: Threshold IMT and traditional physical therapy program
- group B (Active Comparator): twenty ICU-acquired weakness elderly patients will receive chest physiotherapy (cough training, vibration, percussion, rib springing, and postural drainage), 30 minutes of resisted training on upper- and lower-limb muscles (15 min on upper limb and 15 min on lower limb), and 30 minutes of neuromuscular electrical stimulation of lower- and upper-limb muscles (triceps and wrist extensors, dorsiflexors, and quadriceps). sessions will be executed 5 times weekly). The study duration will be 1 month.
  Interventions: Behavioral: traditional physiotherapy program

INTERVENTIONS:
Behavioral: Threshold IMT and traditional physical therapy program — twenty ICU-acquired weakness elderly patients will receive chest physiotherapy (cough training, vibration, percussion, rib springing, and postural drainage), 30 minutes of resisted training on upper- and lower-limb muscles (15 min on upper limb and 15 min on lower limb), and 30 minutes of neuromuscular electrical stimulation of lower- and upper-limb muscles (triceps and wrist extensors, dorsiflexors, and quadriceps). sessions will be executed 5 times weekly). this Group will receive 3-set IMT (two sessions daily via threshold IMT, the set contain 10 repetitions) 5 times weekly. The study duration will be 1 month.
  Arms: group A
Behavioral: traditional physiotherapy program — twenty ICU-acquired weakness elderly patients will receive chest physiotherapy (cough training, vibration, percussion, rib springing, and postural drainage), 30 minutes of resisted training on upper- and lower-limb muscles (15 min on upper limb and 15 min on lower limb), and 30 minutes of neuromuscular electrical stimulation of lower- and upper-limb muscles (triceps and wrist extensors, dorsiflexors, and quadriceps). sessions will be executed 5 times weekly).
  Arms: group B

SUMMARY:
Intensive care unit-acquired weakness (ICU-acquired weakness) may be caused by a variety of different causes. Several studies have shown that ICU-acquired weakness occurs in up to 30% of critically ill patients. It affects daily activities, walking, and functional performance

DETAILED DESCRIPTION:
Forty ICU-acquired weakness elderly patients will be randomly assigned to group A and group B, 20 elderly for each. Both groups will receive chest physiotherapy (cough training, vibration, percussion, rib springing, and postural drainage), 30 minutes of resisted training on upper- and lower-limb muscles (15 min on upper limb and 15 min on lower limb), and 30 minutes of neuromuscular electrical stimulation of lower- and upper-limb muscles (triceps and wrist extensors, dorsiflexors, and quadriceps). sessions will be executed 5 times weekly). Group A only will receive 3-set IMT (two sessions daily via threshold IMT, the set contain 10 repetitions) 5 times weekly. The study duration will be 1 month.

ELIGIBILITY:
Inclusion Criteria:

* sufferers with intensive care unit acquired weakness
* Older sufferers patients with severe walking disability detected by Modified Functional Ambulation Category test,

Exclusion Criteria:

* lower limb amputations
* orthopedic or spinal disc disorders

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 40 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Modified Functional Ambulation Category Test | it will be measured after 1 month
  it is a category test used to assess walking disability

SECONDARY OUTCOMES:
functional vital capacity | It will be measured after 1 month
  the percentage of predicted value of functional vital capacity will be assessed
forced expiatory volume in the first second of expiration | It will be measured after 1 month
  the percentage of predicted value of FEV1 will be assessed
Partial Pressure of Oxygen | It will be measured after 1 month
  it is an arterial blood gas test
Partial Pressure of carbon dioxide | It will be measured after 1 month
  it is an arterial blood gas test
Oxygen saturation | It will be measured after 1 month
  it is an arterial blood gas test
inspiratory muscle strength | It will be measured after 1 month
  it will be measure in cm H2O
expiratory muscle strength | It will be measured after 1 month
  it will be measure in cm H2O
time up and go test | It will be measured after 1 month
  it is time used to walk a three-meter distance
30-second sit to stand | It will be measured after 1 month
  number of (sit to stand) done in 30 seconds
six-minute walk test, | It will be measured after 1 month
  distance walked in 6 minute
10-meter walking test | It will be measured after 1 month
  it is time used to walk a 10-meter distance
mental division of short form 36 | It will be measured after 1 month
  it assess mental component of short form 36 quality of life questionnare
physical division of short form 36 | It will be measured after 1 month
  it assess physical component of short form 36 quality of life questionnare

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo Unoversity, Giza, Egypt

REFERENCES:
- [Derived] Alahmari M, Elsisi HF, Ismail AMA. Functional outcomes of inspiratory muscle training in elderly with intensive care unit-acquired weakness and severe walking disability. Ir J Med Sci. 2025 Apr;194(2):761-769. doi: 10.1007/s11845-025-03876-w. Epub 2025 Feb 3. PMID 39899253